CLINICAL TRIAL: NCT00882869
Title: A Phase 1-2, Open-Label Study of The X-Linked Inhibitor of Apoptosis (XIAP) Antisense AEG35156 in Combination With Sorafenib in Patients With Advanced Hepatocellular Carcinoma (HCC)
Brief Title: XIAP Antisense AEG35156 in Combination With Sorafenib in Patients With Advanced Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aegera Therapeutics (Industry)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Jacques Jolivet, MD, Senior VP Clinical, Aegera Therapeutics Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AEG35156-205
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-07

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Advanced Hepatocellular carcinoma; liver; cancer; antisense; sorafenib
MeSH Terms: conditions — Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AEG35156 antisense IV infusion — Dose escalation (100, 200 and 300 mg/day) over 2 hr infusion, once weekly over 21 days (Day 1, 8, 15)
Drug: Sorafenib — Sorafenib will be administered at 400 mg BID every day
  Other Names: nexavar

SUMMARY:
AEG35156 is a second generation antisense which targets XIAP mRNA to lower XIAP levels and the apoptotic threshold of cancer cells, enhancing their sensitivity to intrinsic death and chemotherapy. Advanced HCC is an attractive target for AEG35156 since XIAP is highly expressed in HCC and may prevent cancer cells from undergoing apoptosis. Second generation antisense molecules are known to accumulate in liver where AEG35156 may down regulate XIAP protein expression in HCC cells thus promoting their apoptotic death.

ELIGIBILITY:
Inclusion Criteria:

* HCC diagnosed by:

  * Histology, or
  * AASLD Criteria in which the diagnosis is made clinically in a patient with a known hepatitis B or cirrhosis of other etiology has a liver mass of > 2cm with typical features of HCC (i.e., hypervascular with washout in the portal/venous phase) on a dynamic imaging study (contrast CT / USG / MRI) or alternatively if the AFP is >200 ng/ml.
* The tumor is not suitable for curative treatment (resection / transplant / local ablative therapies) or the patient is medically inoperable or refuses such treatment.
* At least one measurable lesion according to RECIST criteria.
* Age > 18 years.
* Life expectancy of greater than 12 weeks.
* ECOG performance status ≤ 2 (please refer to Appendix 1).
* Child-Pugh score A or B (please refer to Appendix 2).
* Adequate organ functions defined as:

  * ANC ≥ 1.5 x 109/L
  * Platelet count ≥ 75 x 109/L
  * Creatinine ≤ 1.5 x ULN
  * ALT or AST < 2.5 x ULN
  * Total bilirubin < 50 μmol/L
  * INR <1.7
  * No encephalopathy clinically
  * Normal ECG
* For women of child-producing potential, the use of effective contraceptive methods during the study.
* Prior local therapy to tumor (e.g. surgery, RFA, PEI, chemo-embolization, radiotherapy) is allowed provided that there is a target lesion not subjected to local therapy and/or disease progression has been documented in the target lesion subjected to local therapy. The treatment must be completed at least 4 weeks and patient has recovered from all the acute toxicities of that treatment.
* For patients with hepatitis B, the patient must receive antiviral therapy prior to or with registration.

Exclusion Criteria:

* Child-Pugh score C.
* Patients who have had prior systemic chemotherapy.
* Patients who have had any other cancer related therapy including radiotherapy within 4 weeks prior to entering the study.
* Patients receiving any other investigational agents concurrently.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Patients who have peripheral neuropathy.
* Uncontrolled intercurrent disease such as, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
* Known bleeding diathesis.
* Pregnant or nursing women. NOTE: Women of child-bearing potential must agree to use adequate contraception (sterile or surgically sterile; hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Men who are unwilling to use acceptable forms of birth control when engaging in sexual contact with women of child bearing potential.
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
* Serious nonmalignant disease that could compromise protocol objectives in the opinion of the investigator and/or the sponsor.
* Patients who are currently receiving any other investigational agent. Subjects who have used a previous antisense oligonucleotide in the last 90 days will be excluded.
* Unwillingness or inability to comply with procedures required in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To determine the recommended dose of AEG35156 in combination with sorafenib patients with advanced HCC | 12 months
  13 patients were enrolled into the phase 1 dose escalation part of the study. The recommended dose was determined to be 300 mg.
To evaluate the efficacy of AEG35156 in combination with sorafenib based on PFS(PII) using sorafenib alone for comparison | 12 months

SECONDARY OUTCOMES:
To determine the safety profile of AEG35156 in combination with sorafenib in advanced HCC | 12 months
To determine the response rate of AEG35156 in combination with sorafenib in advanced HCC | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ann Shing Lee, MBChB(CUHK), FHKAM(Rad), Principal Investigator — Tuen Mun Hospital
Locations (3):
- China (3):
  - Tuen Mun Hospital, Tuenmen, New Territories, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong

REFERENCES:
- [Derived] Lee FA, Zee BC, Cheung FY, Kwong P, Chiang CL, Leung KC, Siu SW, Lee C, Lai M, Kwok C, Chong M, Jolivet J, Tung S. Randomized Phase II Study of the X-linked Inhibitor of Apoptosis (XIAP) Antisense AEG35156 in Combination With Sorafenib in Patients With Advanced Hepatocellular Carcinoma (HCC). Am J Clin Oncol. 2016 Dec;39(6):609-613. doi: 10.1097/COC.0000000000000099. PMID 24977690